CLINICAL TRIAL: NCT02384460
Title: A Phase 3, Multi-center, Randomized, Double-Blind, Placebo Controlled Study of the Efficacy and Safety of SD-101 Cream in Patients With Epidermolysis Bullosa
Brief Title: ESSENCE Study: Efficacy and Safety of SD-101 Cream in Participants With Epidermolysis Bullosa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scioderm, Inc. (Industry)
Collaborators: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SD-005; 2014-002288-14 (EudraCT Number); R01-005095-01 (Other: Orphan Product Grant)
Record Dates: First submitted 2015-02-13; First posted 2015-03-10 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Epidermolysis Bullosa
Keywords: Amicus Therapeutics; Scioderm, Inc.; Simplex; Recessive Dystrophic; Junctional non-Herlitz; Epidermolysis Bullosa; SD-101 6%; SD-101-6.0; Allantoin 6%; Zorblisa
MeSH Terms: conditions — Epidermolysis Bullosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SD-101-6.0 cream (Experimental): SD-101-6.0 cream applied topically, once a day to the entire body for a period of 90 days
  Interventions: Drug: SD-101-6.0 cream
- Placebo (SD-101-0.0) cream (Placebo Comparator): SD-101-0.0 (placebo) cream applied topically, once a day to the entire body for a period of 90 days
  Interventions: Drug: Placebo (SD-101-0.0) cream

INTERVENTIONS:
Drug: SD-101-6.0 cream — applied topically once a day for 90 days
  Other Names: SD-101
  Arms: SD-101-6.0 cream
Drug: Placebo (SD-101-0.0) cream — applied topically once a day for 90 days
  Other Names: placebo
  Arms: Placebo (SD-101-0.0) cream

SUMMARY:
The aim was to assess the efficacy and safety of SD-101-6.0 cream versus Placebo (SD-101-0.0) cream in the treatment of skin lesions in participants with Epidermolysis Bullosa. Funding Source - United States Food and Drug Administration (FDA) Office of Orphan Products Development (OOPD).

DETAILED DESCRIPTION:
This was a Phase 3, multi-center, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of SD-101-6.0 cream versus placebo (SD-101-0.0) cream on skin lesions in participants with Simplex, Recessive Dystrophic, or Junctional non-Herlitz Epidermolysis Bullosa. Epidermolysis Bullosa is a rare group of inherited disorders that typically manifest at birth as blistering and lesion formation on the skin in response to little or no apparent trauma. In this study, SD-101-6.0 cream or placebo (SD-101-0.0) cream was to be applied topically, once a day to the entire body for a period of 90 days. Participants had 1 target wound selected at baseline by the investigator. The selected target wound was required to have been present for at least 21 days. Photographic confirmation of the target wound location was collected at baseline, and the picture saved from the first visit was used to confirm location of the target wound at subsequent visits. The participant returned to the study site for Visit 2 (approximately 14 days from baseline), Visit 3 (approximately 30 days from baseline), Visit 4 (approximately 60 days from baseline), and Visit 5 (approximately 90 days from baseline) to have the target wound assessed for the level of healing. In addition, itching, pain, body surface area, target wound closure, and scarring of healed target wound were assessed at each visit. The ARANZ SilhouetteStar™ was used to measure the target wound at all visits.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent form signed by the participant or participant's legal representative; if the participant was under the age of 18 but capable of providing assent, signed assent from the participant.
* Participant (or caretaker) must have been willing to comply with all protocol requirements.
* Diagnosis of Simplex, Recessive Dystrophic, or Junctional non-Herlitz EB.
* Participant must have had 1 target wound (size 10 to 50 cm^2) at study entry.
* Participants 1 month and older.
* Target wound must have been present for at least 21 days.

Exclusion Criteria:

* Participants who did not meet the entry criteria outlined above.
* Selected target wound did not have clinical evidence of local infection.
* Use of any investigational drug within the 30 days before enrollment.
* Use of immunotherapy or cytotoxic chemotherapy within the 60 days before enrollment.
* Use of systemic or topical steroidal therapy within the 30 days before enrollment. (Inhaled steroids and ophthalmic drops containing steroids were allowed).
* Use of systemic antibiotics within the 7 days before enrollment.
* Current or former malignancy.
* Arterial or venous disorder resulting in ulcerated lesions.
* Pregnancy or breastfeeding during the study. (A urine pregnancy test was performed at screening and every 30 days until the final visit for female participants of childbearing potential).
* Females of childbearing potential who were not abstinent and not practicing a medically acceptable method of contraception.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Amicus Therapeutics
Locations (36):
- United States (20):
  - Phoenix, Arizona
  - Redwood City, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Chicago, Illinois
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Hackensack, New Jersey
  - East Setauket, New York
  - New York, New York
  - Chapel Hill, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - San Antonio, Texas
  - Seattle, Washington
- Australia (2):
  - Kogarah, New South Wales
  - Parkville, Victoria
- Salzburg, Austria
- France (3):
  - Nice
  - Paris
  - Toulouse
- Germany (2):
  - Freiburg im Breisgau
  - Hanover
- Tel Aviv, Israel
- Milan, Italy
- Kaunas, Lithuania
- Groningen, Netherlands
- Warsaw, Koszykowa, Poland
- Belgrade, Serbia
- Madrid, Spain
- London, United Kingdom

REFERENCES:
- [Derived] Murrell DF, Paller AS, Bodemer C, Browning J, Nikolic M, Barth JA, Lagast H, Krusinska E, Reha A; ESSENCE Study Group. Wound closure in epidermolysis bullosa: data from the vehicle arm of the phase 3 ESSENCE Study. Orphanet J Rare Dis. 2020 Jul 21;15(1):190. doi: 10.1186/s13023-020-01435-3. PMID 32693833
- [Derived] Paller AS, Browning J, Nikolic M, Bodemer C, Murrell DF, Lenon W, Krusinska E, Reha A, Lagast H, Barth JA; ESSENCE Study Group. Efficacy and tolerability of the investigational topical cream SD-101 (6% allantoin) in patients with epidermolysis bullosa: a phase 3, randomized, double-blind, vehicle-controlled trial (ESSENCE study). Orphanet J Rare Dis. 2020 Jun 23;15(1):158. doi: 10.1186/s13023-020-01419-3. PMID 32576219

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 210 participants screened for this study, 169 participants were randomly assigned, on a 1:1 basis, to treatment with SD-101-6.0 or placebo at 31 study centers in 13 countries. The first participant was enrolled on 11 March 2015 and the last participant completed the study on 05 July 2017.
Pre-assignment Details: Participants had to be >1 month of age with a diagnosis of simplex, recessive dystrophic, or junctional non-Herlitz Epidermolysis Bullosa (EB) and a target wound with a surface area of 10 to 50 cm^2 and ≥21 days old to be considered for participation. Participants who did not meet all inclusion/exclusion criteria were eligible for rescreening.
Groups:
- SD-101-6.0 Cream: Participants applied SD-101-6.0 cream topically, once a day to the entire body for a period of 90 days.
- Placebo (SD-101-0.0) Cream: Participants applied Placebo (SD-101-0.0) cream topically, once a day to the entire body for a period of 90 days.
Period: Overall Study
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream
Started | 82 | 87
Received at Least 1 Dose of Study Drug | 82 | 87
Completed | 75 | 80
Not Completed | 7 | 7
Not completed — Protocol Violation | 0 | 1
Not completed — Returned to previous therapeutic regimen | 0 | 1
Not completed — Adverse Event | 5 | 2
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Elective medical treatment | 1 | 0
Not completed — Non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Placebo (SD-101-0.0) Cream: Placebo (SD-101-0.0) cream applied topically, once a day to the entire body for a period of 90 days.
- Total: Total of all reporting groups
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream | Total
Number analyzed (Participants) | 82 | 87 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (13.15) | 13.9 (13.12) | 13.9 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 48 | 81
  Male | 49 | 39 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 69 | 72 | 141
  Black/African American | 5 | 3 | 8
  Asian | 4 | 8 | 12
  Other | 1 | 1 | 2
  Not Reported | 3 | 3 | 6
EB type [Count of Participants; unit: Participants]
  Simplex | 10 | 8 | 18
  Recessive dystrophic | 57 | 62 | 119
  Junctional non-Herlitz | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Time To Complete Target Wound Closure Within 3 Months
Description: Target wounds were monitored at each study visit for complete closure, defined as skin re-epithelialization without drainage. Time to target wound closure was measured from the date of the first administration of the study drug to the date of target wound closure. Participants were censored if they did not have a response within 3 months, or withdrew earlier before the confirmation of their target wound closing. This primary end point displays the mean time to complete target wound closure, analyzed using a Kaplan-Meier approach.
Time Frame: From baseline to Month 3 visit
Population: ITT population with post-baseline wound closure data and whose target wound had closed within 3 months.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream
Number analyzed (Participants) | 39 | 45
days | 41.6 (25.50) | 53.6 (28.59)
Statistical Analysis 1: Comparison: SD-101-6.0 Cream vs Placebo (SD-101-0.0) Cream; Cox proportional hazards model compares treatment groups with baseline target wound size, target wound age, and EB type as covariates; Test type: Other; p = 0.985, Cox Model Analysis — p-value is for Type 3 chi-square test for comparison between treatments; Hazard Ratio (HR) = 1.004, 95% CI 2-sided [0.651 to 1.549]

2. Primary Outcome: The Percentage Of Participants Experiencing Complete Closure Of Their Target Wound Within 3 Months
Description: Target wounds were monitored at each study visit for complete closure, defined as skin re-epithelialization without drainage. Participants were considered responders if they experienced complete wound closure at the Week 2 or Months 1, 2, or 3 visits. If a target wound was documented to have closed at a given visit, it was considered closed at all subsequent visits. This primary end point displays the percentage of participants from the ITT population who had complete target wound closure by the end of the study period (that is, 3 months). Analysis was performed on participants with post-baseline wound closure data.
Time Frame: From baseline to Month 3 visit
Population: ITT population with post-baseline wound closure data and whose target wound had closed within 3 months.
Measure: Number; unit: percentage of participants
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream
Number analyzed (Participants) | 79 | 84
percentage of participants | 49.4 | 53.6
Statistical Analysis 1: Comparison: SD-101-6.0 Cream vs Placebo (SD-101-0.0) Cream; Comparison between treatment groups of complete closure of target wound within 3 months was performed using a logistic regression model with multiple imputation with EB type, baseline target wound size, and baseline target wound age as covariates; Test type: Other — Multiple imputation was implemented by 2 steps. The first step used Markov Chain Monte Carlo (MCMC) to get monotonic missing data pattern. In the second step, a logistic regression model was used, with the following covariates included in the imputation model: treatment, EB type, baseline target wound size, target wound age, and non-missing data from earlier time points. The seed number was 010005 and the number of imputations was 5; p = 0.39, Regression, Logistic — p-value is from the logistic regression model for treatment comparison; Odds Ratio (OR) = 0.733, 95% CI 2-sided [0.365 to 1.474]

3. Secondary Outcome: Percentage Of Participants Experiencing Complete Closure Of Their Target Wound At Month 1 And Month 2 Visits
Description: Target wounds were monitored at each study visit for complete closure, defined as skin re-epithelialization without drainage. The percentage of participants who completed target wound closure at the Month 1 and Month 2 study visits is displayed. If a target wound was documented to have closed at a given visit, it was considered closed at all subsequent visits.
Time Frame: From baseline to Month 1 and Month 2 visits
Population: Analysis was performed on participants from the ITT population with post-baseline wound closure data.
Measure: Number; unit: percentage of participants
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream
Number analyzed (Participants) | 79 | 84
percentage of participants
  Month 1 | 31.6 | 22.6
  Month 2 | 43.0 | 42.9
Statistical Analysis 1: Comparison: SD-101-6.0 Cream vs Placebo (SD-101-0.0) Cream; Logistic Regression Analysis at Month 1 visit. Comparison between treatment groups of complete closure of target wound within 1 month was performed using a logistic regression model with multiple imputation with EB type, baseline target wound size, and baseline target wound age as covariates; Test type: Other — Multiple imputation was implemented by 2 steps. The first step used MCMC to get the monotonic missing data pattern. In the second step, a logistic regression model was used, with the following covariates included in the imputation method: treatment, EB type, baseline target wound size, target wound age, and non-missing data from earlier time points. The seed number was 01005 and the number of imputations was 5; p = 0.212, Regression, Logistic — p-value is from the logistic regression model for treatment comparison; Odds Ratio (OR) = 1.633, 95% CI 2-sided [0.758 to 3.517]
Statistical Analysis 2: Comparison: SD-101-6.0 Cream vs Placebo (SD-101-0.0) Cream; Logistic Regression Analysis at Month 2 visit. Comparison between treatment groups of complete closure of target wound within 2 months was performed using a logistic regression model with multiple imputation with EB type, baseline target wound size, and baseline target wound age as covariates; Test type: Other — Multiple imputation was implemented by 2 steps. The first step used MCMC to get monotonic missing data pattern. In the second step, a logistic regression model was used, with the following covariates included in the imputation model: treatment, EB type, baseline target wound size, target wound age, and non-missing data from earlier time points. The seed number was 01005 and the number of imputations was 5; p = 0.802, Regression, Logistic — p-value is from the logistic regression model for treatment comparison; Odds Ratio (OR) = 0.891, 95% CI 2-sided [0.436 to 1.821]

4. Secondary Outcome: Change From Baseline In Body Surface Area Index (BSAI) Of Lesional Skin At Month 3 Visit
Description: Lesional skin was defined as areas that contained any of the following: blisters, erosions, ulcerations, scabbing, bullae, or eschars, as well as areas that were weeping, sloughing, oozing, crusted, or denuded. BSAI was calculated as a percentage, ranging from 0% to 100%, of affected body surface area, recorded for each defined body region (that is, head/neck, upper limbs, trunk [includes groin], and lower limbs), multiplied by the weighting factor, then summed for all body regions.
Time Frame: Baseline, Month 3 visit
Population: Analysis was performed on the ITT population. The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage change in BSAI
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream
Number analyzed (Participants) | 75 | 78
Percentage change in BSAI | -4.637 (1.404) | -5.319 (1.354)
Statistical Analysis 1: Comparison: SD-101-6.0 Cream vs Placebo (SD-101-0.0) Cream; Mixed Model Repeated Measures (MMRM) Analysis. The MMRM approach (using restricted maximum likelihood [REML] estimation) was used on each multiply-imputed data set. The model included treatment, baseline BSAI of lesional skin, EB type, visit, and visit-treatment interaction as the fixed effects; Test type: Other — Multiple imputation was used by 2 steps. The first step used MCMC to get monotonic missing data pattern. In the second step, a linear regression model was used, with the following covariates included in the imputation model: treatment, EB type, baseline BSAI of lesional skin, and non-missing data from earlier time points. The seed number was 01005 and the number of imputations was 5; p = 0.706, Mixed Models Analysis — The p-value is calculated based on the hypothesis testing for the difference of least-squares (LS)-means between treatment and placebo; LS means difference = 0.682, 95% CI 2-sided [-2.873 to 4.238]

5. Secondary Outcome: Change From Baseline In BSAI Of Total Body Wound Burden At Month 3 Visit
Description: Total body wound burden was calculated using BSAI. A wound defined as an open area on the skin (that is, epidermal covering disrupted). BSAI was calculated as a percentage, ranging from 0% to 100%, of affected body surface area, recorded for each defined body region (that is, head/neck, upper limbs, lower limbs, trunk [includes groin]), and multiplied by the weighting factor, then summed for all body regions.
Time Frame: Baseline, Month 3 visit
Population: Analysis was performed on the ITT population. The ITT population included all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: Percentage change in BSAI
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream
Number analyzed (Participants) | 75 | 79
Percentage change in BSAI | -3.050 (0.816) | -2.922 (0.813)
Statistical Analysis 1: Comparison: SD-101-6.0 Cream vs Placebo (SD-101-0.0) Cream; MMRM Analysis. The MMRM approach (using REML estimation) was used on each multiply-imputed data set. The model included treatment, baseline BSAI of lesional skin, EB type, visit, and visit-treatment interaction as the fixed effects; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.9, Mixed Models Analysis — The p-value is calculated based on the hypothesis testing for the difference of LS-means between treatment and placebo; LS means difference = 0.128, 95% CI 2-sided [-2.116 to 1.861]

6. Secondary Outcome: Change From Baseline In Itching Score At Day 7
Description: Itching was assessed using the 5-point Itch Man Pruritus Assessment Tool. For participants up to 5 years of age, itching was assessed using caretaker's response and participants 6 years of age and older self-reported their itching assessments based on the following scores: 0=Comfortable, no itch; 1=itches a little, does not interfere with activity; 2=itches more, sometimes interferes with activity; 3=itches a lot, difficult to be still, concentrate; 4=itches most terribly, impossible to sit still or concentrate. Itching scores were categorized into 3 groups based on improvement; Improved or No Itching, Not Improved, and Missing. An itching score reduction from baseline greater than or equal to 1 point on the scale was classed as improved.
Time Frame: Baseline, Day 7
Population: Analysis was performed on the ITT population. The ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream
Number analyzed (Participants) | 77 | 79
units on a scale | -0.5 (1.31) | -0.3 (1.24)
Statistical Analysis 1: Comparison: SD-101-6.0 Cream vs Placebo (SD-101-0.0) Cream; The proportion of participants experiencing improvement in itching versus non-improvement (including missing) was compared between the 2 treatment groups for Day 7 using the logistic regression model with baseline itching score, and EB type as covariates; Test type: Other — Pre-specified; p = 0.262, Regression, Logistic — p-value is from the logistic regression model for treatment comparison; Odds Ratio (OR) = 1.445, 95% CI 2-sided [0.759 to 2.752]

7. Secondary Outcome: Change From Baseline In Pain Score At Day 7
Description: Change in pain assessed at Day 7 compared to baseline was measured using the Face, Legs, Activity, Cry, and Consolability (FLACC) behavioral scale for participants 1 month to 3 years of age. Each of the 5 FLACC categories was scored from 0 to 2, which resulted in a total score between 0 and 10 with 0=Relaxed and comfortable, 1 to 3=Mild discomfort, 4 to 6=Moderate pain, and 7 to 10=Severe discomfort/pain. For participants 4 years of age and older, the "Wong Faces Pain Scale" was used. This scale shows a series of faces ranging from a happy face at 0, which represents "no hurt," to a crying face at 10, which represents "hurts worst". Pain scores were categorized into 3 groups based on improvement: Improved or No Pain, Not Improved, and Missing. A pain score reduction from baseline greater than or equal to 2 points on the scale was classed as improved.
Time Frame: Baseline, Day 7
Population: Analysis was performed on the ITT population. The ITT population included all randomized participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream
Number analyzed (Participants) | 77 | 80
units on a scale | -0.3 (2.57) | -0.6 (3.07)
Statistical Analysis 1: Comparison: SD-101-6.0 Cream vs Placebo (SD-101-0.0) Cream; The proportion of participants experiencing improvement in pain versus non-improvement (including missing) was compared between the 2 treatment groups for Day 7 using the logistic regression model with baseline pain score and EB type as covariates; Test type: Other — Pre-specified; p = 0.098, Regression, Logistic — p-value is from the logistic regression model for treatment comparison; Odds Ratio (OR) = 0.596, 95% CI 2-sided [0.323 to 1.1]

ADVERSE EVENTS:
Time Frame: From baseline up to 3 months.
Description: Adverse events (AEs) were defined as treatment-emergent AEs if the AE occurred on or after the first date of application of study drug.
Arm/Group | SD-101-6.0 Cream | Placebo (SD-101-0.0) Cream
All-Cause Mortality (participants affected / at risk) | 0/82 | 1/87
Serious Adverse Events (participants affected / at risk) | 4/82 | 8/87
Other Adverse Events (participants affected / at risk) | 49/82 | 46/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SD-101-6.0 Cream (N=82) | Placebo (SD-101-0.0) Cream (N=87)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Cystitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 2
Staphylococcal skin infection (Infections and infestations) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Aggression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SD-101-6.0 Cream (N=82) | Placebo (SD-101-0.0) Cream (N=87)
Anemia (Blood and lymphatic system disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2
Pain (General disorders) | 1 | 4
Pyrexia (General disorders) | 5 | 9
Ear infection (Infections and infestations) | 1 | 4
Nasopharyngitis (Infections and infestations) | 11 | 3
Pharyngitis (Infections and infestations) | 1 | 4
Skin bacterial infection (Infections and infestations) | 1 | 4
Skin infection (Infections and infestations) | 3 | 9
Staphyloccocal skin infection (Infections and infestations) | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 4 | 9
Wound infection (Infections and infestations) | 6 | 5
Wound infection staphylococcal (Infections and infestations) | 1 | 4
Fall (Injury, poisoning and procedural complications) | 3 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Blister (Skin and subcutaneous tissue disorders) | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 8
Rash (Skin and subcutaneous tissue disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT02384460/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT02384460/SAP_001.pdf